CLINICAL TRIAL: NCT04542174
Title: Prospective Non-Interventional Post Market Clinical Follow-up Study TRJ® - 8 Years Results
Brief Title: PMCF 8 Year Results TRJ®
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1908
Record Dates: First submitted 2020-09-02; First posted 2020-09-09 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Arthroplasty, Replacement, Hip; Follow-Up Study
Keywords: Trochanter retaining joint replacement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The intention of this Post Market Clinical Follow-Up study is to obtain mid-term results of the TRJ® endoprosthesis. Aim is to include those patients that have received a TRJ® Total Hip Arthroplasty in 2012 and already did participated in a clinical study taking place in 2014 to obtain 2 years results

ELIGIBILITY:
Inclusion Criteria:

* patients have received a TRJ® prosthesis in 2012
* Patient did participate in the 2 years results evaluation 2014
* Patient gave his written consent for study participation

Exclusion Criteria:

* patient is pregnant
* patient < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-09-26 (Actual); Study Completion 2021-09-26 (Actual)

PRIMARY OUTCOMES:
Survival rate of the stem | at follow-up examination approximately 8 years after primary intervention
  The survival of the TRJ® stem prosthesis will be analyzed using the "Kaplan-Meier". Isolated revisions of the inlay and / or of the acetabular components (with the stem being kept in place) are documented, but assessed separately.

SECONDARY OUTCOMES:
Hip Dysfunction and Osteoarthritis Outcome Score (HOOS) | at follow-up examination approximately 8 years after primary intervention
  The Hip Dysfunction and Osteoarthritis Outcome Score (HOOS) is a 40 items patient reported outcome score (PROM) designed specifically to evaluate the physical functionality of hip osteoarthritis patients. The HOOS offers 5 subgroups, each with 100 points as best result.
Harris Hip Score (HHS) | at follow-up examination approximately 8 years after primary intervention
  The Harris Hip Score (HHS) is one of the most used scores in total hip arthroplasty, mainly combining range of motion questions with questions regarding daily life activities.
Rate of Adverse and Serious Adverse Events | at follow-up examination approximately 8 years after primary intervention
  All Adverse Events (AE) / Serious Adverse Events (SAE) either observed during the follow-up examination, found in the patient file of the hospital or reported by the patient will be documented. Only those AE and SAE that could be related to the investigational product or the TRJ® Total Hip Arthroplasty procedure in 2012 are of interest.
Pain Assessment | at follow-up examination approximately 8 years after primary intervention
  Pain will be measured with a Visual Analogue Scale (VAS), at rest and when walking on flat ground. The Visual Analog Scale (VAS) is a 10 cm line with anchor statements on the left (no pain) and on the right (extreme pain). The patient is asked to mark their current pain level on the line.
Radiological Outcome: Inlay wear | at follow-up examination approximately 8 years after primary intervention
  Inlay wear is assessed on AP x-rays of the cup and will be analysed according to the zones defined by DeLee and Charnley. "Charnley" and "Gruen" zones of the hip are distinct zones used in assessment of aseptic loosening in total hip joint replacements.
Radiological Outcome: Bony Osseointegration or conspicuous features of the cup | at follow-up examination approximately 8 years after primary intervention
  Bony Osseointegration or conspicuous features of the Cup are assessed on anterior-posterior x-rays of the cup and will be analysed according to the zones defined by DeLee and Charnley. "Charnley" and "Gruen" zones of the hip are distinct zones used in assessment of aseptic loosening in total hip joint replacements.
Radiological Outcome: Migration of the stem in mm | at follow-up examination approximately 8 years after primary intervention
  Migration of the stem is assessed in [mm] relative to discharge x-rays
Radiological Outcome: Bone resorption at the medial stem neck | at follow-up examination approximately 8 years after primary intervention
  Bone Resorption is assessed on anterior-posterior and lateral x-rays of the stem
Radiological Outcome: Bone resorption at the Trochanter Major | at follow-up examination approximately 8 years after primary intervention
  Bone Resorption is assessed on anterior-posterior and lateral x-rays of the stem
Radiological Outcome: Evaluation of bony osseointegration or conspicuous features of the stem | at follow-up examination approximately 8 years after primary intervention
  Bony Osseointegration or conspicuous features of the stem are assessed on anterior-posterior and lateral x-rays of the stem and will be analysed according to the zones defined by Gruen. "Charnley" and "Gruen" zones of the hip are distinct zones used in assessment of aseptic loosening in total hip joint replacements
Radiological Outcome: Heterotopic Ossification | at follow-up examination approximately 8 years after primary intervention
  Brooker classification divides heterotopic ossifications that form following total hip replacement to four classes. Class I: islands of bone within soft tissues around hip; Class II: bone spurs in pelvis or proximal end of femur leaving ≥1 cm between the opposing bone surfaces; Class III: bone spurs that extend from pelvis or the proximal end of femur, which reduce the space between the opposing bone surfaces to <1cm; Class IV: ankylosis of the hip on x-ray

CONTACTS AND LOCATIONS:
Locations (1):
- Dreifaltigkeitskrankenhaus Köln, Cologne, Germany